CLINICAL TRIAL: NCT00452361
Title: A Randomized, Open-label, Comparative Evaluation of Conversion From Calcineurin Inhibitors to Sirolimus Versus Continued Use of Calcineurin Inhibitors in Renal Allograft Recipient
Brief Title: Study Evaluating of Calcineurin Inhibitors Versus Sirolimus in Renal Allograft Recipient
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H-101864
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-07

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sirolimus therapy
  Interventions: Drug: Sirolimus+MMF or MPS or AZA+Steroid
- 2 (Active Comparator): Calcineurin Inhibitor therapy (either cyclosporine or tacrolimus)
  Interventions: Drug: Calcineurin Inhibitors (either cyclosporine or tacrolimus)+MMF or MPS or AZA+Steroid

INTERVENTIONS:
Drug: Sirolimus+MMF or MPS or AZA+Steroid — Corticosteroids will be administered according to local practice, within a daily maintenance dosage range of 2.5 to15 mg for prednisone or prednisolone (2 to 12 mg/day for methylprednisolone) or the alternate day equivalent.
  Arms: 1
Drug: Calcineurin Inhibitors (either cyclosporine or tacrolimus)+MMF or MPS or AZA+Steroid — The maintenance dose of:
  1. MMF will not exceed 1500 mg/day or PMS will not exceed 1080 mg/day
  2. AZA will not exceed 75 mg/day
  Thereafter, at the discretion of the investigator, MMF/MPS or AZA may be:
  1. continued for the entire 104-week period of randomized therapy
  2. subsequently discontinued
  3. restarted after discontinuation
  Arms: 2

SUMMARY:
This study will evaluate whether conversion from cyclosporine, a calcineurin inhibitor (CI) to sirolimus (SRL) results in improved long-term renal function without a negative impact on safety or immunosuppressive efficacy, and to further examine the potential of SRL to reduce the severity and/or progression of chronic allograft nephropathy (CAN).

DETAILED DESCRIPTION:
This open-label, randomized, parallel-group, comparative, outpatient study will be conducted in multiple centers in Taiwan.

The study will randomize approximately 120 patients. 80 patients will be randomized to the SRL therapy group (conversion from CI- to SRL-based immunosuppression: group A) and 40 patients to the CI therapy group (continued CI therapy: group B).

Dosage and Administration

SRL Therapy: At the time of randomization on day 1, each patient will have been receiving:

* triple therapy with a CI (tacrolimus or CsA) that began at the time of transplantation or within 2 weeks thereafter AND
* corticosteroids corresponding to a dosage range of 2.5 to 15 mg/day for prednisone or prednisolone (2 to 12 mg/day for methylprednisolone) or the alternate day equivalent for at least 12 weeks before randomization, PLUS
* either MMF (minimum dose 500 mg/day)/MPS (minimum dose 360 mg/day) or AZA (minimum dose 50 mg/day) for at least 12 weeks before randomization.

SRL will be added to the immunosuppressive regimen for Group A. Group B will continue on this CI immunosuppressive regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age.
* Subjects who are 6 to 60 months after renal transplantation.
* Subjects who have a stable graft function.

Exclusion Criteria:

* Subjects with active major infection, including HIV, decreased platelets, elevated lipids, or multiple organ transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Select Cities, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in Taiwan from April 2007 to May 2008.
Pre-assignment Details: After consent and eligibility criteria patients needed to be receiving: triple therapy with a Calcineurin Inhibitor (CI) (tacrolimus or cyclosporine) that began at the time of transplantation or ≤2 weeks thereafter and corticosteroids plus either mycophenolate mofetil (MMF)/mycophenolate sodium (MPS) or azathioprine (AZA) for at least 12 weeks.
Groups:
- Sirolimus (SRL): SRL added to the immunosuppressive regimen at a daily maintenance dose of 2 mg, following a loading dose of 6 mg. The dose of SRL adjusted as necessary to maintain a whole blood trough concentration range of 10 to 15 ng/mL. CI dose was reduced by 50% and discontinued within 2 weeks if SRL at the target trough level. Once SRL trough level was at target range, MMF dose reduced to a maximum of 1500 mg/day or MPS dose reduced to a maximum of 1080 mg/day and AZA dose reduced to a maximum of 75 mg/day. Corticosteroids were administered according to local practice, within a daily maintenance dosage range (2.5 to 15 mg for prednisone or prednisolone; 2 to 12 mg/day for methylprednisolone) or the alternate day equivalent.
- Calcineurin Inhibitor (CI): Patients will continue to receive a CI (tacrolimus or CsA). At the discretion of the investigator, patients will be permitted to: (a) change from MMF/MPS to AZA or vice versa, and from CsA to tacrolimus or vice versa; (b) continue MMF/MPS or AZA for the entire 104-week period of randomized therapy; or (c) discontinue MMF/MPS or AZA and subsequently restart either one after discontinuation. Whole blood CsA or tacrolimus trough concentrations will be monitored at designated intervals and the CI dose adjusted to maintain the following trough concentration ranges: CsA 50-250 ng/mL and Tacrolimus 4-10 ng/mL.
Period: Overall Study
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Started | 21 | 10
Completed | 0 | 0
Not Completed | 21 | 10
Not completed — Adverse Event | 8 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Premature termination | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI) | Total
Number analyzed (Participants) | 21 | 10 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 46.8 (7.9) | 42.2 (13.9) | 43.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 13
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Glomerular Filtration Rate (GFR) Change From Baseline
Description: GFR is an index of kidney function. GFR describes the flow rate of filtered fluid through the kidney. GFR can be measured directly or estimated using established formulas. GFR was calculated using Nankivell formula. A normal GFR is > 90 mL/min, although children and older people usually have a lower GFR. Lower values indicate poor kidney function. A GFR <15 is consistent with kidney failure.
Time Frame: 104 weeks
Population: No patients completed 104 weeks and therefore no data were available for efficacy analysis.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Glomerular Filtration Rate (GFR)
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Glomerular Filtration Rate (GFR)
Description: as for outcome 1
Time Frame: Baseline and Week 52
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Glomerular Filtration Rate (GFR)
Description: as for outcome 1
Time Frame: Baseline and Week 104
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patient and Graft Survival
Description: Patient survival defined as participants living with or without a functioning graft. Graft survival defined as those participants who did not experience graft loss. Graft loss defined as physical loss (nephrectomy), functional loss (necessitating maintenance dialysis for >8 weeks), retransplant or death during the first 12 months after randomization.
Time Frame: Week 24
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient and Graft Survival
Description: as for outcome 5
Time Frame: Week 52
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Patient and Graft Survival
Description: as for outcome 5
Time Frame: Week 104
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 24
Description: Value at Week 24 minus value at baseline.
Time Frame: Baseline and Week 24
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 52
Description: Value at Week 52 minus value at baseline.
Time Frame: Baseline and Week 52
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 104
Description: Value at Week 104 minus value at baseline.
Time Frame: Baseline and Week 104
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 24
Description: Value at Week 24 minus value at baseline.
Time Frame: Baseline and Week 24
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 52
Description: Value at Week 52 minus value at baseline.
Time Frame: Baseline and Week 52
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 104
Description: Value at Week 104 minus value at baseline.
Time Frame: Baseline and Week 104
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in the Severity and Progression of Biopsy-Confirmed Chronic Allograft Nephropathy (CAN) at Week 104
Time Frame: Baseline and Week 104
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Occurence of Acute Rejection or Premature Withdrawal From Study Medication for Any Reason by Week 52
Time Frame: Weeks 52
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Occurence of Acute Rejection or Premature Withdrawal From Study Medication for Any Reason by Week 104
Time Frame: Week 104
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Incidence and Severity of Biopsy-Confirmed Acute Rejection at Week 24
Time Frame: Week 24
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Incidence and Severity of Biopsy-Confirmed Acute Rejection at Week 52
Time Frame: Week 52
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Incidence and Severity of Biopsy-Confirmed Acute Rejection at Week 104
Time Frame: Week 104
Population: Insufficient or no data available for efficacy analyses because study was terminated early.
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sirolimus (SRL) | Calcineurin Inhibitor (CI)
Serious Adverse Events (participants affected / at risk) | 6/21 | 2/10
Other Adverse Events (participants affected / at risk) | 78/21 | 18/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (SRL) (N=21) | Calcineurin Inhibitor (CI) (N=10)
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cellulitis (General disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lens dislocation (Eye disorders) | 0 | 1
Appendicitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (SRL) (N=21) | Calcineurin Inhibitor (CI) (N=10)
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Eyelid oedema (Eye disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 11 | 2
Tooth ache (Gastrointestinal disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Herpes virus infection (General disorders) | 2 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Aspartate aminotransferase increased (Investigations) | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Dizziness (Nervous system disorders) | 2 | 0
Insomina (Nervous system disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Epistaxis (Blood and lymphatic system disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 8 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Study terminated early due to difficulties in enrolling qualified patients. No patients completed 104 weeks (primary outcome); a few completed 60 weeks. Insufficient data were available for efficacy analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.